CLINICAL TRIAL: NCT01033851
Title: Stress Reduction Techniques and Anxiety: Therapeutic and Neuroendocrine Effects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Elizabeth A. Hoge, MD, Assistant Psychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-P-000275; 5K23AT004432 (NIH)
Record Dates: First submitted 2009-12-09; First posted 2009-12-17 (Estimated); Results first posted 2013-06-11 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness Based Stress Reduction (Active Comparator): Mindfulness Based Stress Reduction (MBSR) is an 8-week group intervention that trains participants in mindfulness meditation techniques.
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Stress Management Education (Active Comparator): Stress Management Education (SME) is an 8-week group intervention that educates participants about stress physiology and health lifestyle changes.
  Interventions: Behavioral: Stress Management Education

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — 8 week course
  Arms: Mindfulness Based Stress Reduction
Behavioral: Stress Management Education — 8 week course
  Arms: Stress Management Education

SUMMARY:
Current therapies for Generalized Anxiety Disorder (GAD) have limited effectiveness. This study measures the efficacy of two different approaches to reducing anxiety and stress. One approach uses education, nutrition, exercise, and time management training, and another uses mindfulness meditation and yoga, which is taught as part of the Mindfulness-based stress reduction (MBSR) course, an 8-week manualized mindfulness intervention. We hypothesize that the two approaches will reduce anxiety in individuals with GAD in different ways. We will measure changes in stress hormones associated with these changes.

ELIGIBILITY:
Inclusion Criteria:

* Adults with generalized anxiety disorder
* medically healthy

Exclusion Criteria:

* substance abuse
* history of other psychiatric diagnoses such as psychosis, Obsessive Compulsive Disorder, PTSD
* use of certain types of psychotherapy, meditation training, yoga
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-03; Primary Completion 2012-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Hoge, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Hoge EA, Guidos BM, Mete M, Bui E, Pollack MH, Simon NM, Dutton MA. Effects of mindfulness meditation on occupational functioning and health care utilization in individuals with anxiety. J Psychosom Res. 2017 Apr;95:7-11. doi: 10.1016/j.jpsychores.2017.01.011. Epub 2017 Jan 23. PMID 28314552
- [Derived] Hoge EA, Bui E, Marques L, Metcalf CA, Morris LK, Robinaugh DJ, Worthington JJ, Pollack MH, Simon NM. Randomized controlled trial of mindfulness meditation for generalized anxiety disorder: effects on anxiety and stress reactivity. J Clin Psychiatry. 2013 Aug;74(8):786-92. doi: 10.4088/JCP.12m08083. PMID 23541163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by media advertisement and referral between December 2008 and February 2011.
Groups:
- Mindfulness Based Stress Reduction; Stress Management Education: Weekly 2 hour class, given for 8 weeks total.
Period: Overall Study
Arm/Group | Mindfulness Based Stress Reduction | Stress Management Education
Started | 48 | 41
Completed | 45 | 34
Not Completed | 3 | 7
Not completed — Withdrawal by Subject | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Stress Reduction | Stress Management Education | Total
Number analyzed (Participants) | 48 | 41 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 40 | 84
  >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (14) | 37 (12) | 39 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 25 | 19 | 44
Region of Enrollment [Number; unit: participants]
  United States | 48 | 41 | 89

OUTCOME MEASURES:

1. Primary Outcome: Active Symptoms of Generalized Anxiety Disorder
Description: The Hamilton Anxiety Scale (HAMA) was defined as the primary anxiety outcome variable. This scale has 14 items describing symptoms of anxiety, each answered on a 0-4 scale, with 0 for a single question generally representing no symptoms, and 4 representing severe levels of the symptom. The total score is calculated by adding all the items together, for a possible total score of 0 to 56.
Time Frame: 2 months
Population: The population analyzed included all participants who attended at least one class of an intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Based Stress Reduction | Stress Management Education
Number analyzed (Participants) | 48 | 41
units on a scale | 13.65 (7.01) | 16.27 (7.26)

2. Secondary Outcome: Clinical Global Impression of Severity (CGIS) of Anxiety Symptoms.
Description: This is an overal clinical measure of anxiety symptoms after examining and interviewing the patient. The scale is one global item, that scores from 1 (1= not ill at all) to 7 (7= among the most extremely ill).
Time Frame: 2 months
Population: The population analyzed included all participants attending at least one class of an intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Based Stress Reduction | Stress Management Education
Number analyzed (Participants) | 48 | 41
units on a scale | 3.15 (1.11) | 3.58 (1.28)
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Stress Management Education; A repeated measure ANOVA, with time as the repeated measure, treatment arm as between-subjects factor and CGI-S score as the dependent variable, found a main effect of time (F(1,84)=62.19, p<0.001) and a significant treatment arm X time interaction (F(1,84)=4.51, p=0.0366); Test type: Superiority or Other; p = 0.0366, ANOVA

ADVERSE EVENTS:
Time Frame: 2 months
Description: A validated questionnaire was used to assess adverse events.
Arm/Group | Mindfulness Based Stress Reduction | Stress Management Education
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/41
Other Adverse Events (participants affected / at risk) | 1/48 | 1/41
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Based Stress Reduction (N=48) | Stress Management Education (N=41)
muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
sleep disruption (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No